CLINICAL TRIAL: NCT01166698
Title: A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group, 2-part Study to Assess the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Inhaled Doses of AZD9819 in Healthy Subjects
Brief Title: Single Centre, Double-blind, Single and Multiple Ascending Inhaled Doses of AZD9819 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D3020C00001
Record Dates: First submitted 2010-07-20; First posted 2010-07-21 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Healthy Volunteers; Safety; Tolerability
Keywords: Safety; tolerability; healthy; inhalation
MeSH Terms: conditions — Respiratory Aspiration | interventions — AZD9819

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD9819 (Experimental): Inhaled suspension
  Interventions: Drug: AZD9819
- Placebo (Placebo Comparator): Inhaled suspension
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD9819 — Inhaled single doses of suspension via SPIRA nebuliser
  Arms: AZD9819
Drug: AZD9819 — Inhaled multiple doses of suspension via SPIRA nebuliser, once daily for 10 (maximum 14) days
  Other Names: Part B (multiple ascending doses)
  Arms: AZD9819
Drug: Placebo — Inhaled doses of suspension via SPIRA nebuliser given either as single (Part A) or multiple doses (Part B)
  Other Names: Part A and B
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess safety and tolerability of AZD9819 following inhaled administration of single and multiple increasing doses, and to estimate the maximum dose that is tolerated in healthy people.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Healthy male and female (non-child bearing potential) subjects aged 18 to 50 years with suitable veins for cannulation or repeated venepuncture.
* Have a body mass index (BMI) between 18 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg

Exclusion Criteria:

* Any clinically significant disease or disorder
* Any clinically significant abnormalities at screening examination
* Use of any prescribed or non-prescribed medication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Safety variables (ECG variables, adverse events, blood pressure, pulse, body temp, safety lab) | Frequent safety measurements during the study from screening period to follow-up

SECONDARY OUTCOMES:
Pharmacokinetic variables of AZD9819 by assessment of drug concentrations in plasma | Multiple PK blood samples from pre-dose until 96 hours post last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, London, United Kingdom